CLINICAL TRIAL: NCT02411656
Title: A Phase II Study of Anti-PD-1 (MK-3475) Therapy in Patients With Metastatic Inflammatory Breast Cancer (IBC) or Non-IBC Triple Negative Breast Cancer (TNBC) Who Have Achieved Clinical Response or Stable Disease to Prior Chemotherapy
Brief Title: Pembrolizumab in Treating Patients With Stage IV Metastatic or Recurrent Inflammatory Breast Cancer or Triple-Negative Breast Cancer Who Have Achieved Clinical Response or Stable Disease to Prior Chemotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0533; NCI-2015-00671 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0533 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Results first posted 2025-07-02 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Edema; Erythema; Estrogen Receptor Negative; HER2/Neu Negative; Peau d'Orange; Progesterone Receptor Negative; Recurrent Inflammatory Breast Carcinoma; Stage IV Inflammatory Breast Carcinoma; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Edema; Erythema; Inflammatory Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab 200mg IV over approximately 30 minutes on day 1. Cycles repeat every 21 days for 8 cycles and then pembrolizumab 400mg IV every 42 days for total up to 24 months in the absence of disease progression or unacceptable toxicity
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab works in treating patients with stage IV inflammatory breast cancer or triple-negative breast cancer that has spread to other places in the body (metastatic) or has come back (recurrent), and who have achieved clinical response or stable disease to prior chemotherapy. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Primary Objective: To assess the efficacy of MK-3475 as a single agent in patients with metastatic IBC or non-IBC TNBC

EXPLORATORY OBJECTIVES:

1. To investigate the association between biomarkers in the peripheral blood and tumor tissue, such as PD-L1 expression, with safety and efficacy for IBC or non-IBC TNBC patients treated with MK-3475.
2. To determine the disease control rate of metastatic IBC or non-IBC TNBC patients who have achieved clinical response or stable disease to the systemic therapy.
3. To investigate the association between biomarkers and efficacy by RNA-sequencing of exosomes in blood and tumor for IBC or non-IBC TNBC patients treated with MK-3475.
4. To investigate the 5-year OS for IBC or non-IBC TNBC patients treated with MK-3475

OUTLINE:

Patients receive pembrolizumab 200mg IV over approximately 30 minutes on day 1. Cycles repeat every 21 days for 8 cycles and then pembrolizumab 400mg IV every 42 days for total up to 24 months in the absence of disease progression or unacceptable toxicity

After completion of study treatment, patients are followed up at approximately 1 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Is willing and able to provide written informed consent for the trial
* Is a female or male and >/= 18 years of age
* Has histological confirmation of HER2 normal breast carcinoma with a clinical diagnosis of IBC based on presence of inflammatory changes in the involved breast, including diffuse erythema and edema (peau d'orange), with or without an underlying palpable mass involving the majority of the skin of the breast; pathological evidence of dermal lymphatic invasion should be noted but is not required for diagnosis of inflammatory breast cancer regardless estrogen receptor (ER)/progesterone receptor (PR) status; OR has histological confirmation of triple negative breast carcinoma (HER2 normal, ER/PR < 10%) without clinical diagnosis of IBC
* Has stage IV or recurrent disease that has been treated
* Has clinical response or stable disease for minimum of two months (three cycles of every three week chemotherapy or 8 weeks of weekly regimen, etc.) after receiving any prior chemotherapy for metastatic/recurrent disease; a minimum of two cycles (6-8 weeks) of chemotherapy is required to determine clinical response.

Per RECIST criteria 1.1, Clinical response for measurable disease is defined as complete response (CR) or partial response (PR); for non-measurable disease only (i.e. bone metastasis, ascites, pleural effusion, and pathological lymph nodes >/= 10 to <15 mm short axis) is defined as persistence of one or more non-target lesion(s) and no increase in overall tumor burden.

* Is HER2 normal, defined as HER2 0 or 1+ by IHC and negative by FISH if performed; or HER2 is 2+ by IHC and negative by FISH; or HER2 negative by FISH if IHC is not performed.
* Has a performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Has adequate organ function as determined by the following laboratory values:

ANC >/= 1000 /mcL, Platelets >/=100,000 /mcL, Hgb >/= 9 g/dL, creatinine levels < 1.5 x ULN, Total bilirubin </= 1.5 x ULN, ALT and AST </= 2.5 x ULN or </=5 x ULN for participants with liver metastases.

* Participants of childbearing potential should be willing to use effective methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through at least 4 months after the last dose of study drug. Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year. Effective methods of birth control include 1). Use of hormonal birth control methods: pills, shots/injections, implants (placed under the skin by a health care provider), or patches (placed on the skin); 2).Intrauterine devices (IUDs); 3).Using 2 barrier methods (each partner must use 1 barrier method) with a spermicide. Males must use the male condom (latex or other synthetic material) with spermicide. Females must choose either a Diaphragm with spermicide, or Cervical cap with spermicide, or a sponge (spermicide is already in the contraceptive sponge).
* Has negative serum or urine pregnancy test for participants of childbearing potential

Exclusion Criteria:

* Is currently participating in a study of an investigational anti-cancer agent
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy
* Has not recovered from adverse events due to prior therapies, i.e. monoclonal antibody, chemotherapy, targeted small molecule therapy, radiation therapy, or surgery. (Note: Participants with ≤ grade 2 neuropathy, alopecia and general disorders and administration site conditions [per Common Terminology Criteria for Adverse Events (CTCAE version 4.0) are an exception to this criterion and may qualify for the study)
* Has a known malignancy (other than breast cancer) except basal cell carcinoma or squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; participants with previously treated brain metastases may participate if they are stable, and have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; participants with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Participants that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Participants with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has an active infection requiring systemic therapy
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Has a known history of human immunodeficiency virus (HIV)
* Has a known active hepatitis B or hepatitis C
* Have received a live vaccine within 30 days prior to the first dose of trial treatment
* Is receiving concurrent anti-cancer therapy for metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2028-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bora Lim, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Pembrolizumab): Pembrolizumab 200mg IV every 21 days for 8 cycles and then 400mg IV every 42 days for total up to 24 months in the absence of disease progression or unacceptable toxicity
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab)
Started | 45
Completed | 8
Not Completed | 37
Not completed — Adverse Event | 4
Not completed — Clinical Progression | 33

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 54 [34 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 38
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Efficacy of Pembrolizumab as a Single Agent in Patients With Metastatic IBC or Non-IBC TNBC
Description: The disease control rate (DCR) was assessed. The DCR was defined as the proportion of all treated patients with a lack of progression within 4 months as determined by radiologic imaging or clinical assessment.
Time Frame: 4 months from the start of therapy
Population: Patients who received a total of at least 2 cycles of pembrolizumab were analyzed. Two patients were excluded because they discontinued the study treatment due to toxicity after one dose.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 43
percentage of participants | 58.1

2. Other Pre Specified Outcome: Correlation Between PD-L1 IHC Status and Overall Survival in Patients Treated With Pembrolizumab
Description: PD-L1 satus in tumor tissue was determined by IHC analysis: positive CPS≥ 10, negative CPS <10. Median OS and 95% confidence interval are estimated by the PD-L1 status in tumor tissue (positive vs. negative).
Time Frame: From the first dose of pembrolizumab up to 5 years
Population: The patients with tumor samples available
Measure: Median (95% Confidence Interval); unit: months
Groups:
- PD-L1 Negative: Patients with PD-L1 CPS <10 based on IHC analysis
- PD-L1 Positive: Patients with PD-L1 CPS ≥10 based on IHC analysis
Arm/Group | PD-L1 Negative | PD-L1 Positive
Number analyzed (Participants) | 20 | 12
months | 26.0 [13.3 to 55.9] | 31.9 [9.2 to NA] — The upper bound of the 95% CI for the median overall survival (OS) was not estimable due to the high proportion of censored observations and insufficient number of events beyond the median, limiting the precision of upper-tail estimation.

3. Other Pre Specified Outcome: Correlation Between PD-L1 IHC Status and Progression-Free Survival in Patients Treated With Pembrolizumab
Description: PD-L1 expression in tumor tissue was assessed by immunohistochemistry (IHC), with CPS ≥10 defined as PD-L1 positive and CPS <10 as PD-L1 negative.Median PFS and 95% confidence interval are estimated by the PD-L1 status in tumor tissue (positive vs. negative).
Time Frame: From the first dose of pembrolizumab up to 3 years
Population: The patients with tumor samples available
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PD-L1 Negative | PD-L1 Positive
Number analyzed (Participants) | 20 | 12
months | 3.9 [2.5 to 6.5] | 5.7 [3.4 to NA] — The upper bound of the 95% CI for the median overall survival (OS) was not estimable due to the high proportion of censored observations and insufficient number of events beyond the median, limiting the precision of upper-tail estimation.

4. Other Pre Specified Outcome: To Investigate the Association Between Biomarkers and Efficacy by RNA-sequencing of Exosomes in Blood and Tumor for IBC or Non-IBC TNBC Patients Treated With Pembrolizumab.
Description: RNA-sequencing will be performed with RNA extracted from plasma at baseline.
Time Frame: Baseline
Population: No data is available. As a result, no participants were included in this outcome measure analysis.
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Overall Survival for IBC or Non-IBC TNBC Patients Treated With Pembrolizumab
Description: Overall survival time from the registration date was estimated using Kaplan-Meier method.
Time Frame: From registration date to up to 5 years
Population: Patients who received a total of at least 2 cycles of pembrolizumab were analyzed.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 43
years | 2.17 [1.11 to 3.19]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was assessed through study completion, up to 5 years; all Adverse Events were collected from the time of the first protocol-specific intervention until 3 months after the last dose of drug, up to 3 years
Description: Adverse events were assessed according to the CTCAE version 4.0. All study patients who had received any dose of Pembrolizumab were evaluable for safety. Unexpected adverse events, including laboratory adverse events deemed clinically significant by the investigator, were graded and recorded.
Arm/Group | Treatment (Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 34/45
Serious Adverse Events (participants affected / at risk) | 13/45
Other Adverse Events (participants affected / at risk) | 40/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Pembrolizumab) (N=45)
Abdominal pain (Gastrointestinal disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Optic Neuritis (Eye disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Gait disturbance (General disorders) | 1
Headache (Nervous system disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Infection (Infections and infestations) | 2
Infusion related reaction (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Skin infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Pembrolizumab) (N=45)
Abdominal pain (Gastrointestinal disorders) | 6
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 6
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 4
Anemia (Blood and lymphatic system disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 4
Anxiety (Psychiatric disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Aspartate aminotransferase increased (Investigations) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5
Breast pain (Reproductive system and breast disorders) | 3
Bruising (Injury, poisoning and procedural complications) | 4
Heart Rate increased (Cardiac disorders) | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3
Chills (General disorders) | 3
Constipation (Gastrointestinal disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Creatinine increased (Investigations) | 3
Diarrhea (Gastrointestinal disorders) | 13
Dizziness (Nervous system disorders) | 5
Dry eye (Eye disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 5
Dysgeusia (Nervous system disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10
Edema limbs (General disorders) | 4
TSH decreased (Endocrine disorders) | 3
Fall (Injury, poisoning and procedural complications) | 3
Fatigue (General disorders) | 18
Fever (General disorders) | 4
Flu like symptoms (General disorders) | 3
Gait disturbance (General disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5
Headache (Nervous system disorders) | 19
Hot flashes (Vascular disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypertension (Vascular disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypothyroidism (Endocrine disorders) | 7
Upper respiratory infection (Infections and infestations) | 4
Insomnia (Psychiatric disorders) | 6
Lactate dehydrogenase (LDH) increased (Investigations) | 4
Lymphedema (Vascular disorders) | 3
Lymphocyte count decreased (Investigations) | 4
Memory impairment (Nervous system disorders) | 3
Hyperphosphatemia (Metabolism and nutrition disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 5
Muscle cramps (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 16
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12
Nausea (Gastrointestinal disorders) | 20
Pain (General disorders) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Paresthesia (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash acneiform (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 15
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6
Stomach pain (Gastrointestinal disorders) | 4
Upper respiratory infection (Infections and infestations) | 6
Vomiting (Gastrointestinal disorders) | 15
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT02411656/Prot_SAP_000.pdf